CLINICAL TRIAL: NCT04860947
Title: Assessment of Serum Neurofilament-light Chain (NfL) and Glial Fibrillary Acidic Protein (GFAP) Levels, Atrophy of the Macular Ganglion Cell Complex (GCC) by Optical Coherence Tomography (OCT) and Whole Brain Atrophy by MRI to Predict Evolution of Neurological Disability in Multiple Sclerosis Patients
Brief Title: Assessment of NfL and GFAP Levels, Atrophy of the Macula GCC by OCT and Whole Brain Atrophy by MRI to Predict Evolution of Neurological Disability in MS Patients
Acronym: NFL OCT
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Institut de Recherches en Biothérapie (Unknown)
Responsible Party: Sponsor
Other Study IDs: CIVI/2018/ET-01; 2018-A03152-53 (Other: ANSM)
Record Dates: First submitted 2021-04-16; First posted 2021-04-27 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis
Keywords: GFAP; NfL
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MS patients
  Interventions: Diagnostic Test: Brain MRI; Diagnostic Test: Spinal Cord MRI; Diagnostic Test: Retinal imaging

INTERVENTIONS:
Diagnostic Test: Brain MRI — * Axial DWI with ADC card
  * Axial 2D TSE T2/DP or 3DT2
  * Gadolinium injection (0.1 mmol/kg)
  * 3D Fluid-attenuated inversion recovery
  * 3D T1 with Gadolinium injection.
Diagnostic Test: Spinal Cord MRI — Sagittal T2 Sagittal T1 with Gadolinium injection
Diagnostic Test: Retinal imaging — spectral-domain high definition optical coherence tomography

SUMMARY:
The investigators hypothesize that serum neurofilament-light chain (NfL) levels at baseline and decrease of the macular ganglion cell complex (GCC) thickness at one year vs. baseline are as good as progression of whole brain atrophy at one year vs. baseline to predict later evolution of neurological disability in multiple sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been correctly informed.
* The patient must have given their informed and signed consent.
* The patient must be insured or beneficiary of a health insurance plan.
* The patient is at least (≥)18 years old.
* The patient has experienced a CIS, has currently a RRMS or progressive MS with:

  * Less than 10 years of disease duration;
  * With or without DMD;
  * EDSS score 0 - 7.0.

Exclusion Criteria:

* The patient is in an exclusion period determined by a previous study.
* The patient is under judicial protection.
* The patient refuses to sign the consent.
* It is impossible to correctly inform the patient (Inability to understand the study, language problem).
* The patient is pregnant or breast-feeding.
* Patient has a bilateral optic neuritis or other significant ophthalmological antecedent.
* Patient with MRI contra-indications.
* patient has a contraindication to gadolinium injection
* The patient has bilateral optic neuritis or other significant ophthalmological antecedent
* Patient is having a relapse or has had a relapse in the last 3 months
* The patient has a severe psychiatric illness
* The patient has severe chronic alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of consecutive adult patients, of both sexes, recruited during consultations for a CIS, RRMS or progressive MS at the Neurology department of Nîmes University Hospital (CHU). The patients recruited will have an EDSS score comprised between 0 - 7.0.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in serum Neurofilament Light Chain serum levels since baseline | Baseline; 1 year
  pg/mL; measured by digital ELISA
Change in serum Glial Fibrillary Acidic Protein (GFAP) serum levels since baseline | Baseline; 1 year
  pg/mL; measured by digital ELISA
Change in Ganglion Cell Complex thickness since baseline | Baseline; 1 year
  Measured by Optical Coherence Tomography
Change in whole brain volume since baseline | Baseline; 1 year
  Assessed by MRI
Expanded Disability Status Scale | Baseline
  Eight functional systems scored on a scale of 0 (no disability) to 5 or 6 (more severe disability)
Expanded Disability Status Scale | 3 years
  Eight functional systems scored on a scale of 0 (no disability) to 5 or 6 (more severe disability)

SECONDARY OUTCOMES:
Whole brain volume | Inclusion
  assessed by MRI
Whole brain volume | 6 Months
  assessed by MRI
Whole brain volume | 1 Year
  assessed by MRI
Whole brain volume | 2 years
  assessed by MRI
Whole brain volume | 3 Years
  assessed by MRI
Whole brain volume | 4 Years
  assessed by MRI
Whole brain volume | 5 years
  assessed by MRI
Whole brain volume | any relapse (max 5 years)
  assessed by MRI
Expanded Disability Status Scale | Inclusion
  Eight functional systems scored on a scale of 0 (no disability) to 5 or 6 (more severe disability)
Expanded Disability Status Scale | 6 Months
  Eight functional systems scored on a scale of 0 (no disability) to 5 or 6 (more severe disability)
Expanded Disability Status Scale | 1 year
  Eight functional systems scored on a scale of 0 (no disability) to 5 or 6 (more severe disability)
Expanded Disability Status Scale | 18 months
  Eight functional systems scored on a scale of 0 (no disability) to 5 or 6 (more severe disability)
Expanded Disability Status Scale | 2 years
  Eight functional systems scored on a scale of 0 (no disability) to 5 or 6 (more severe disability)
Expanded Disability Status Scale | 2.5 years
  Eight functional systems scored on a scale of 0 (no disability) to 5 or 6 (more severe disability)
Expanded Disability Status Scale | 3 years
  Eight functional systems scored on a scale of 0 (no disability) to 5 or 6 (more severe disability)
Expanded Disability Status Scale | 3.5 years
  Eight functional systems scored on a scale of 0 (no disability) to 5 or 6 (more severe disability)
Expanded Disability Status Scale | 4 years
  Eight functional systems scored on a scale of 0 (no disability) to 5 or 6 (more severe disability)
Expanded Disability Status Scale | 4.5 years
  Eight functional systems scored on a scale of 0 (no disability) to 5 or 6 (more severe disability)
Expanded Disability Status Scale | 5 years
  Eight functional systems scored on a scale of 0 (no disability) to 5 or 6 (more severe disability)
Expanded Disability Status Scale | Any relapse (Maximum 5 years)
  Eight functional systems scored on a scale of 0 (no disability) to 5 or 6 (more severe disability)
Peripapillary Retinal Nerve Fibre Layer atrophy and Ganglion Cell Complex thickness | Inclusion
  assessed by Optical Coherence Tomography
Peripapillary Retinal Nerve Fibre Layer atrophy and Ganglion Cell Complex thickness | 6 Months
  assessed by Optical Coherence Tomography
Peripapillary Retinal Nerve Fibre Layer atrophy and Ganglion Cell Complex thickness | 1 Year
  assessed by Optical Coherence Tomography
Peripapillary Retinal Nerve Fibre Layer atrophy and Ganglion Cell Complex thickness | 18 Months
  assessed by Optical Coherence Tomography
Peripapillary Retinal Nerve Fibre Layer atrophy and Ganglion Cell Complex thickness | 2 years
  assessed by Optical Coherence Tomography
Peripapillary Retinal Nerve Fibre Layer atrophy and Ganglion Cell Complex thickness | 3 Years
  assessed by Optical Coherence Tomography
Peripapillary Retinal Nerve Fibre Layer atrophy and Ganglion Cell Complex thickness | 4 Years
  assessed by Optical Coherence Tomography
Peripapillary Retinal Nerve Fibre Layer atrophy and Ganglion Cell Complex thickness | 5 Years
  assessed by Optical Coherence Tomography
Peripapillary Retinal Nerve Fibre Layer atrophy and Ganglion Cell Complex thickness | Any relapse (maximum 5 Years)
  assessed by Optical Coherence Tomography
Gadolinium-enhanced lesions | Inclusion
  assessed by MRI
Gadolinium-enhanced lesions | 6 Months
  assessed by MRI
Gadolinium-enhanced lesions | 1 Year
  assessed by MRI
Gadolinium-enhanced lesions | 2 years
  assessed by MRI
Gadolinium-enhanced lesions | 3 Years
  assessed by MRI
Gadolinium-enhanced lesions | 4 Years
  assessed by MRI
Gadolinium-enhanced lesions | 5 Years
  assessed by MRI
Gadolinium-enhanced lesions | Any relapse (Maximum 5 Years)
  assessed by MRI
T2 lesion volume, | Inclusion
  assessed by MRI
T2 lesion volume, | 6 Months
  assessed by MRI
T2 lesion volume, | 1 Year
  assessed by MRI
T2 lesion volume, | 2 years
  assessed by MRI
T2 lesion volume, | 3 Years
  assessed by MRI
T2 lesion volume, | 4 Years
  assessed by MRI
T2 lesion volume, | 5 years
  assessed by MRI
T2 lesion volume, | Any relapse (maximum 5 years)
  assessed by MRI
Grey matter atrophy | Inclusion
  assessed by MRI
Grey matter atrophy | 6 Months
  assessed by MRI
Grey matter atrophy | 1 Year
  assessed by MRI
Grey matter atrophy | 2 years
  assessed by MRI
Grey matter atrophy | 3 Years
  assessed by MRI
Grey matter atrophy | 4 Years
  assessed by MRI
Grey matter atrophy | 5 Years
  assessed by MRI
Grey matter atrophy | Any relapse (maximum 5 Years)
  assessed by MRI
White matter atrophy | Inclusion
  assessed by MRI
White matter atrophy | 6 Months
  assessed by MRI
White matter atrophy | 1 Year
  assessed by MRI
White matter atrophy | 2 years
  assessed by MRI
White matter atrophy | 3 Years
  assessed by MRI
White matter atrophy | 4 Years
  assessed by MRI
White matter atrophy | 5 years
  assessed by MRI
White matter atrophy | Any relapse (maximum 5 years)
  assessed by MRI
Thalamic atrophy | Inclusion
  assessed by MRI
Thalamic atrophy | 6 Months
  assessed by MRI
Thalamic atrophy | 1 Year
  assessed by MRI
Thalamic atrophy | 2 years
  assessed by MRI
Thalamic atrophy | 3 Years
  assessed by MRI
Thalamic atrophy | 4 Years
  assessed by MRI
Thalamic atrophy | 5 years
  assessed by MRI
Thalamic atrophy | Any relapse (maximum 5 years)
  assessed by MRI
Disease modifying drugs classification | Inclusion
  Drug class (1st, 2nd or 3rd line)
Disease modifying drugs classification | until end of study (5 years)
  Drug class (1st, 2nd or 3rd line)
serum NfL levels | 6 Months
  pg/mL; measured by digital ELISA
serum GFAP levels | 6 Months
  pg/mL; measured by digital ELISA
serum NfL levels | 2 years
  pg/mL; measured by digital ELISA
serum GFAP levels | 2 years
  pg/mL; measured by digital ELISA
serum NfL levels | 3 years
  pg/mL; measured by digital ELISA
serum GFAP levels | 3 years
  pg/mL; measured by digital ELISA
serum NfL levels | 4 years
  pg/mL; measured by digital ELISA
serum GFAP levels | 4 years
  pg/mL; measured by digital ELISA
serum NfL levels | 5 years
  pg/mL; measured by digital ELISA
serum GFAP levels | 5 years
  pg/mL; measured by digital ELISA
serum NfL levels | Any relapse (maximum 5 years)
  pg/mL; measured by digital ELISA
serum GFAP levels | Any relapse (maximum 5 years)
  pg/mL; measured by digital ELISA
Multiple Sclerosis Functional Composite | Inclusion
  21-item test that includes 3 different functional subtests: the timed 25-Foot Walk, the 9-Hole Peg Test and the Paced Auditory Serial Addition Test (PASAT)
Multiple Sclerosis Functional Composite | 6 Months
  21-item test that includes 3 different functional subtests: the timed 25-Foot Walk, the 9-Hole Peg Test and the Paced Auditory Serial Addition Test (PASAT)
Multiple Sclerosis Functional Composite | 1 Year
  21-item test that includes 3 different functional subtests: the timed 25-Foot Walk, the 9-Hole Peg Test and the Paced Auditory Serial Addition Test (PASAT)
Multiple Sclerosis Functional Composite | 2 years
  21-item test that includes 3 different functional subtests: the timed 25-Foot Walk, the 9-Hole Peg Test and the Paced Auditory Serial Addition Test (PASAT)
Multiple Sclerosis Functional Composite | 3 years
  21-item test that includes 3 different functional subtests: the timed 25-Foot Walk, the 9-Hole Peg Test and the Paced Auditory Serial Addition Test (PASAT)
Multiple Sclerosis Functional Composite | 4 years
  21-item test that includes 3 different functional subtests: the timed 25-Foot Walk, the 9-Hole Peg Test and the Paced Auditory Serial Addition Test (PASAT)
Multiple Sclerosis Functional Composite | 5 years
  21-item test that includes 3 different functional subtests: the timed 25-Foot Walk, the 9-Hole Peg Test and the Paced Auditory Serial Addition Test (PASAT)
Multiple Sclerosis Functional Composite | Any relapse (maximum 5 years)
  21-item test that includes 3 different functional subtests: the timed 25-Foot Walk, the 9-Hole Peg Test and the Paced Auditory Serial Addition Test (PASAT)
Time to walk 100 meters | Inclusion
  Seconds
Time to walk 100 meters | 6 Months
  Seconds
Time to walk 100 meters | 1 Year
  Seconds
Time to walk 100 meters | 2 years
  Seconds
Time to walk 100 meters | 3 years
  Seconds
Time to walk 100 meters | 4 years
  Seconds
Time to walk 100 meters | 5 years
  Seconds
Time to walk 100 meters | Any relapse (maximum 5 years)
  Seconds
2 Minute walking distance | Inclusion
  Meters
2 Minute walking distance | 6 Months
  Meters
2 Minute walking distance | 1 Year
  Meters
2 Minute walking distance | 2 years
  Meters
2 Minute walking distance | 3 years
  Meters
2 Minute walking distance | 4 years
  Meters
2 Minute walking distance | 5 years
  Meters
2 Minute walking distance | Any relapse (maximum 5 years)
  Meters
Cognitive Impairment | Inclusion
  Symbol Digit Modalities Test
Cognitive Impairment | 6 months
  Symbol Digit Modalities Test
Cognitive Impairment | 1 Year
  Symbol Digit Modalities Test
Cognitive Impairment | 2 years
  Symbol Digit Modalities Test
Cognitive Impairment | 3 years
  Symbol Digit Modalities Test
Cognitive Impairment | 4 years
  Symbol Digit Modalities Test
Cognitive Impairment | 5 years
  Symbol Digit Modalities Test
Cognitive Impairment | Any relapse (maximum 5 years)
  Symbol Digit Modalities Test
Cognitive evaluation | Inclusion
  Brief International Cognitive Assessment for Multiple Sclerosis
Cognitive evaluation | 6 Months
  Brief International Cognitive Assessment for Multiple Sclerosis
Cognitive evaluation | 1 Year
  Brief International Cognitive Assessment for Multiple Sclerosis
Cognitive evaluation | 2 years
  Brief International Cognitive Assessment for Multiple Sclerosis
Cognitive evaluation | 3 years
  Brief International Cognitive Assessment for Multiple Sclerosis
Cognitive evaluation | 4 years
  Brief International Cognitive Assessment for Multiple Sclerosis
Cognitive evaluation | 5 years
  Brief International Cognitive Assessment for Multiple Sclerosis
Cognitive evaluation | Any relapse (maximum 5 years)
  Brief International Cognitive Assessment for Multiple Sclerosis
Health-related quality of life | Inclusion
  EQ-5D-5L
Health-related quality of life | 6 Months
  EQ-5D-5L
Health-related quality of life | 1 Year
  EQ-5D-5L
Health-related quality of life | 2 years
  EQ-5D-5L
Health-related quality of life | 3 years
  EQ-5D-5L
Health-related quality of life | 4 years
  EQ-5D-5L
Health-related quality of life | 5 years
  EQ-5D-5L
Health-related quality of life | Any relapse (maximum 5 years)
  EQ-5D-5L
Impact of MS on daily life | Inclusion
  Multiple Sclerosis Impact Scale (MSIS-29)
Impact of MS on daily life | 6 Months
  Multiple Sclerosis Impact Scale (MSIS-29)
Impact of MS on daily life | 1 Year
  Multiple Sclerosis Impact Scale (MSIS-29)
Impact of MS on daily life | 2 years
  Multiple Sclerosis Impact Scale (MSIS-29)
Impact of MS on daily life | 3 years
  Multiple Sclerosis Impact Scale (MSIS-29)
Impact of MS on daily life | 4 years
  Multiple Sclerosis Impact Scale (MSIS-29)
Impact of MS on daily life | 5 years
  Multiple Sclerosis Impact Scale (MSIS-29)
Impact of MS on daily life | Any relapse (maximum 5 years)
  Multiple Sclerosis Impact Scale (MSIS-29)
Fatigue | Inclusion
  Modified Fatigue Impact Scale
Fatigue | 6 Months
  Modified Fatigue Impact Scale
Fatigue | 1 Year
  Modified Fatigue Impact Scale
Fatigue | 2 years
  Modified Fatigue Impact Scale
Fatigue | 3 years
  Modified Fatigue Impact Scale
Fatigue | 4 years
  Modified Fatigue Impact Scale
Fatigue | 5 years
  Modified Fatigue Impact Scale
Fatigue | Any relapse (maximum 5 years)
  Modified Fatigue Impact Scale
Visual acuity | Inclusion
  0= low, 10= good
Visual acuity | 6 Months
  0= low, 10= good
Visual acuity | 1 Year
  0= low, 10= good
Visual acuity | 2 years
  0= low, 10= good
Visual acuity | 3 years
  0= low, 10= good
Visual acuity | 4 years
  0= low, 10= good
Visual acuity | 5 years
  0= low, 10= good
Visual acuity | Any relapse (maximum 5 years)
  0= low, 10 good
Low contrast visual acuity | Inclusion
  0= low, 10 good
Low contrast visual acuity | 6 Months
  0= low, 10 good
Low contrast visual acuity | 1 Year
  0= low, 10 good
Low contrast visual acuity | 2 years
  0= low, 10 good
Low contrast visual acuity | 3 years,
  0= low, 10 good
Low contrast visual acuity | 4 years
  0= low, 10 good
Low contrast visual acuity | 5 years
  0= low, 10 good
Low contrast visual acuity | Any relapse (maximum 5 years)
  0= low, 10 good
Relapse description | At relapse (maximum 5 years)
  monofocal, plurifocal
Number of new lesions | At relapse (maximum 5 years)
  Measured by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Eric Thouvenot, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France